CLINICAL TRIAL: NCT03631940
Title: Umbilical Cord Milking in Non-Vigorous Infants
Acronym: MINVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Sharp Mary Birch Hospital for Women & Newborns (Other); Sharp Grossmont Hospital (Other); University of Utah (Other); University of Alberta (Other); Poznan University of Medical Sciences (Other); IWK Health Centre (Other); University of California, Davis (Other); Loma Linda University (Other); George Washington University (Other); Providence Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director, Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MINVI; 5R01HD096023-02 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Birth Asphyxia
Keywords: Umbilical Cord Milking; Immediate Cord Clamping; Resuscitation
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Experimental): The delivering practitioner will place the newborn below the level of the incision (at the edge of the table) at C/S and a second team member will milk the cord four times. For vaginal delivery, the delivering obstetrician, midwife or perinatal provider will hold the infant against their body or place the infant on the mother's abdomen and the cord will be milked either four times by the obstetrical provider or by a second team member. For the cord milking procedure, the obstetrical provider will milk the entire length of umbilical cord over two seconds, repeating three additional times as described previously. This time is not significantly different from the time for ECC as we have demonstrated in our previous trials.
  Interventions: Procedure: Umbilical Cord Milking
- Early Cord Clamping (Active Comparator): This will occur by clamping the umbilical cord as soon as possible. Since both ECC and UCM will occur after a brief assessment, it is important to note that the cord clamping time will be longer than in previously conducted preterm trials (average 20 seconds) which performed the intervention on all subjects regardless of whether or not they were vigorous. In all cases, the cord clamping time will be documented to ensure consistency.
  Interventions: Procedure: Early Cord Clamping

INTERVENTIONS:
Procedure: Umbilical Cord Milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 15-20 seconds.
  Arms: Umbilical Cord Milking
Procedure: Early Cord Clamping — The umbilical cord is clamped within 60 seconds of delivery.
  Arms: Early Cord Clamping

SUMMARY:
The investigators will conduct a study of non-vigorous term infants to determine if umbilical cord milking (UCM) results in a lower rate of NICU admissions than early clamping and cutting of the umbilical cord at birth for infants who need resuscitation.

DETAILED DESCRIPTION:
At birth, it is critical that an infant begins breathing quickly. The infant has to switch from relying on the placenta for oxygen to using its lungs for the first time. The currently recommended practice for infants who need resuscitation is to immediately clamp the umbilical cord. Animal studies show that clamping the cord before the baby breathes can cause the heart beat to slow and can decrease the amount of blood being pumped out of the heart each minute. This study will test whether infants will benefit from UCM. The cord will be quickly milked four times before cutting and will not delay the resuscitation procedures. This study is important because when there is need for resuscitation, neither UCM or delayed cord clamping, are recommended by national and international organizations due to lack of evidence. Yet, several large studies from around the world have identified that infants needing resuscitation are more likely to develop conditions such as cerebral palsy, autism and other developmental problems.

The trial is a cluster crossover design in which each hospital will be randomly assigned to use either early cord clamping or UCM for any infant needing resuscitation over a period of 12 months. Then sites will change to the other method for an additional 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-vigorous newborns born between 35-42 weeks gestation

Exclusion Criteria:

* Known major congenital or chromosomal anomalies of newborn
* Known cardiac defects other than small ASD, VSD and PDA
* Complete placental abruption/cutting through the placenta at time of delivery
* Monochorionic multiples
* Cord anomaly (i.e. cord avulsion, true knot)
* Presence of non-reducible nuchal cord
* Perinatal providers unaware of the protocol
* Incomplete delivery data
* Infants born in extremis, for whom additional treatment will not be offered

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1730 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (10):
- United States (7):
  - University of California, Davis, Davis, California
  - Loma Linda Medical Center, Loma Linda, California
  - Sharp Grossmont Hospital, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - George Washington University, Washington D.C., District of Columbia
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Utah/IMH, Salt Lake City, Utah
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Dalhousie, New Brunswick
- Poznan University of Medical Science, Poznan, Poland

REFERENCES:
- [Derived] Katheria AC, El Ghormli L, Clark E, Yoder B, Schmolzer GM, Law BHY, El-Naggar W, Rittenberg D, Sheth S, Martin C, Vora F, Lakshminrusimha S, Underwood M, Mazela J, Kaempf J, Tomlinson M, Gollin Y, Rich W, Morales A, Varner M, Poeltler D, Vaucher Y, Mercer J, Finer N, Rice MM. Two-Year Outcomes of Umbilical Cord Milking in Nonvigorous Infants: A Secondary Analysis of the MINVI Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2416870. doi: 10.1001/jamanetworkopen.2024.16870. PMID 38949814
- See also: MINVI NIRS Substudy — http://clinicaltrials.gov/ct2/show/NCT03621956
- See also: MINVI Follow-up study — https://clinicaltrials.gov/ct2/show/NCT03621943
- See also: MINVI Echocardiogram Substudy — https://clinicaltrials.gov/ct2/show/NCT03798093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 sites were randomized to perform umbilical cord milking or early cord clamping for eligible neonate-mother dyads. Research staff at each sites approached eligible neonate-mother dyads after delivery for written informed consent for additional data collection. Hospital recruited neonate-mother dyads in the initial period from January 2019 to January 2020 and from February 2020 and May 2021 for the crossover period. Neonate-mother dyads participated in a single period of the study.
Pre-assignment Details: Prior to the initiation of recruitment each participating hospital was assigned to perform umbilical cord milking or early cord clamping on non-vigorous neonates-mother dyads delivered during the recruitment period.
  Prior to the start of recruitment in the crossover study period (Study Period 2) a 1-2-month washout period was specified by the protocol for the purpose of site hospital staff retraining and to assess adherence to the new assigned intervention.
Units Other Than Participants: Hospitals
Groups:
- Umbilical Cord Milking, Then Early Cord Clamping - Neonate-Mother Dyad: Umbilical Cord Milking performed in the initial phase and Early Cord Clamping performed in the crossover phase.
- Early Cord Clamping, Then Umbilical Cord Milking - Neonate-Mother Dyad: Early Cord Clamping was performed in the initial phase and Umbilical Cord Milking in the crossover phase
Period: Initial Randomized Intervention Period 1
Arm/Group | Umbilical Cord Milking, Then Early Cord Clamping - Neonate-Mother Dyad | Early Cord Clamping, Then Umbilical Cord Milking - Neonate-Mother Dyad
Started (In the initial period, ten sites were randomized to perform either umbilical cord milking or early cord clamping for all neonates meeting inclusion criteria and born during the participating hospitals' study recruitment period.) | 366; 5 Hospitals (Five hospitals assigned to perform umbilical cord milking on all neonates meeting eligibility criteria and born during the hospital's initial recruitment period. 366 participants enrolled from sites randomized to perform umbilical cord milking in the initial recruitment period) | 494; 5 Hospitals (Five hospitals assigned to perform early cord clamping on all neonates meeting eligibility criteria and born during the hospital's initial recruitment period. 494 participants were enrolled from sites randomized to perform early cord clamping in the initial recruitment period)
Completed | 366; 5 Hospitals (Five hospitals reached their enrollment goal during the initial recruitment period. Participants: 366 neonates meet eligibility criteria and delivered at a participating hospital assigned to perform umbilical cord milking during the initial recruitment period and neonate's disposition following resuscitation in the delivery room was collected.) | 494; 5 Hospitals (Five hospitals reached their enrollment goal during the initial recruitment period. Participants: 494 neonates meet eligibility criteria and delivered at a participating hospital assigned to perform umbilical cord milking during the initial recruitment period and neonate's disposition following resuscitation in the delivery room was collected.)
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Crossover Intervention Period 2
Arm/Group | Umbilical Cord Milking, Then Early Cord Clamping - Neonate-Mother Dyad | Early Cord Clamping, Then Umbilical Cord Milking - Neonate-Mother Dyad
Started (Crossover involved the Hospitals changing the assigned procedure performed for neonates who met eligibility criteria during the participating hospital's crossover recruitment period. Because the procedure (umbilical cord management at the time of delivery) can only be performed once per neonate the counts of participants in the crossover period are independent from the initial period.) | 364; 5 Hospitals (Five hospitals assigned to perform early cord clamping on all neonates meeting eligibility criteria and born during the hospital's crossover recruitment period. 364 participants were enrolled from sites randomized to perform early cord clamping in the crossover recruitment period.) | 506; 5 Hospitals (Five hospitals assigned to perform early cord clamping on all neonates meeting eligibility criteria and born during the hospital's crossover recruitment period. 506 participants enrolled from sites randomized to perform umbilical cord milking in the crossover recruitment period.)
Completed | 364; 5 Hospitals (Five hospitals reached their enrollment goal during the crossover recruitment period. Participants: 364 neonates meet eligibility criteria and delivered at a participating hospital assigned to perform early cord clamping during the crossover recruitment period and neonate's disposition following resuscitation in the delivery room was collected.) | 506; 5 Hospitals (Five hospitals reached their enrollment goal during the crossover recruitment period. Participants: 506 neonates meet eligibility criteria and delivered at a participating hospital assigned to perform umbilical cord milking during the crossover recruitment period and neonate's disposition following resuscitation in the delivery room was collected.)
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals

BASELINE CHARACTERISTICS:
Population: Baseline data was collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval. Maternal sex and region of enrollment were not collected.
Groups:
- Umbilical Cord Milking - Neonate: All neonates who received umbilical cord milking intervention at the time of birth.
  Umbilical Cord Milking: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping - Neonate: All neonates who received early cord clamping at the time of birth. Early Cord Clamping: The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate | Total
Number analyzed (Participants) | 872 | 858 | 1730
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Infant gestational age at birth reported in weeks.
  weeks
    Infants gestational age at birth | 39.3 [38.1 to 40.3] | 39.4 [38.1 to 40.3] | 39.3 [38.1 to 40.3]
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Maternal age at the time of delivery reported in years Population: Baseline data including maternal age was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  years
    Maternal age at time of delivery: number analyzed (Participants) | 606 | 612 | 1218
    Maternal age at time of delivery | 31 [27 to 35] | 30 [27 to 35] | 31 [27 to 35]
Sex: Female, Male [Count of Participants; unit: Participants] — Infant sex: Female, Males Population: Baseline data including neonatal sex was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval. Maternal sex was not collected.
  Participants
    Neonatal Sex: number analyzed (Participants) | 835 | 810 | 1645
    Neonatal Sex: Female | 375 | 355 | 730
    Neonatal Sex: Male | 460 | 455 | 915
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Neonatal ethnicity as reported by birth parent.
  Participants
    Neonatal Ethnicity: Hispanic or Latino | 113 | 152 | 265
    Neonatal Ethnicity: Not Hispanic or Latino | 460 | 379 | 839
    Neonatal Ethnicity: Unknown or Not Reported | 299 | 327 | 626
Race (NIH/OMB) [Count of Participants; unit: Participants] — Neonatal race as reported by birth parent.
  Participants
    Neonatal Race: American Indian or Alaska Native | 9 | 5 | 14
    Neonatal Race: Asian | 39 | 45 | 84
    Neonatal Race: Native Hawaiian or Other Pacific Islander | 2 | 7 | 9
    Neonatal Race: Black or African American | 50 | 47 | 97
    Neonatal Race: White | 333 | 320 | 653
    Neonatal Race: More than one race | 102 | 107 | 209
    Neonatal Race: Unknown or Not Reported | 337 | 327 | 664
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported maternal race and ethnicity.
  Participants
    Non-Hispanic Black Mother | 55 | 53 | 108
    Non-Hispanic Asian Mother | 49 | 56 | 105
    Non-Hispanic White Mother | 338 | 303 | 641
    Non-Hispanic Native American Mother | 14 | 5 | 19
    Non-Hispanic Pacific Islander Mother | 6 | 9 | 15
    Non-Hispanic Multiracial Mother | 16 | 22 | 38
    Maternal ethnicity/race not stated or unknown | 297 | 274 | 571
    Hispanic Mother | 97 | 136 | 233
Region of Enrollment [Number; unit: neonate participants] — Region of enrollment determined based on neonate's birth hospital location.
  neonate participants
    Canada | 227 | 228 | 455
    United States | 625 | 602 | 1227
    Poland | 20 | 28 | 48
Maternal age [Median (Inter-Quartile Range); unit: years] | 31 [27 to 35] | 30 [27 to 35] | 31 [27 to 35]
Maternal level of education: some college education [Count of Participants; unit: Participants] — Self-reported maternal level of education of at least some college education or higher degree. Population: Baseline data including level of education was only collected from participants who provided written consent for additional data collection. Disclosure of level of education was voluntary and not disclosed by all participants.
  Participants
    number analyzed (Participants) | 536 | 508 | 1044
    (all) | 404 | 384 | 788
Maternal hypertension [Count of Participants; unit: Participants] — Number of neonates delivered by a mother who experienced hypertension during pregnancy. Population: Baseline data including maternal hypertension status was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  Participants
    number analyzed (Participants) | 757 | 727 | 1484
    (all) | 154 | 118 | 272
Maternal diabetes [Count of Participants; unit: Participants] — Number of neonates delivered by a mother with diabetes during pregnancy. Population: Baseline data including maternal diabetes status was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  Participants
    number analyzed (Participants) | 757 | 727 | 1484
    (all) | 106 | 92 | 198
Maternal intrauterine inflammation or infection [Count of Participants; unit: Participants] — Number of neonates delivered by a mother diagnosed with intrauterine inflammation or intrauterine infection. Population: Baseline data including maternal intrauterine inflammation or infection status was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  Participants
    number analyzed (Participants) | 757 | 728 | 1485
    (all) | 84 | 96 | 180
Maternal group B streptococcus infection [Count of Participants; unit: Participants] — Number of neonates delivered by a mother with a positive group B streptococcus culture. Population: Baseline data including maternal group B streptococcus infection status was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  Participants
    number analyzed (Participants) | 756 | 728 | 1484
    (all) | 164 | 139 | 303
Number of hours membranes were ruptured before delivery of neonate [Median (Inter-Quartile Range); unit: hours] — Population: Baseline data including length of rupture of membranes was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  hours
    number analyzed (Participants) | 752 | 719 | 1471
    (all) | 7 [1 to 14] | 6 [1 to 14] | 6 [1 to 14]
Maternal general anesthesia [Count of Participants; unit: Participants] — Number of neonates delivered by a mother who was administered general anesthesia at the time of delivery. Population: Baseline data including general anesthesia was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  Participants
    number analyzed (Participants) | 606 | 612 | 1218
    (all) | 41 | 41 | 82
Multiple gestation birth [Count of Participants; unit: Participants] — Number of neonates delivered by a mother with a multiple gestation pregnancy Population: Baseline data including multiple gestation status was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  Participants
    number analyzed (Participants) | 752 | 730 | 1482
    (all) | 21 | 29 | 50
Maternal narcotic or central nervous system depressant medication ≤ 2 hours before delivery [Count of Participants; unit: Participants] — Number of neonates delivered by a mother who was administered an intravenous/oral narcotic or central nervous system depressant medication within 2 hours before delivery.
  Participants | 63 | 66 | 129
Mode of delivery [Count of Participants; unit: Participants] — Method used to deliver neonate.
  Participants
    Vaginal | 395 | 397 | 792
    Cesarean | 362 | 321 | 683
    Unknown | 115 | 140 | 255
Neonatal birth weight [Median (Inter-Quartile Range); unit: grams] — Population: Baseline data including neonatal birthweight was only collected from participants who provided written consent for additional data collection or via waiver of consent for sites with ethics board approval.
  grams
    number analyzed (Participants) | 757 | 730 | 1487
    (all) | 3355 [300 to 3705] | 3395 [2960 to 3775] | 3370 [2985 to 3750]

OUTCOME MEASURES:

1. Primary Outcome: Number of Neonatal Participants Admitted to the NICU for Predefined Criteria
Description: Number of neonatal participants admitted to the neonatal intensive care unit for study-specific predefined criteria including respiratory distress, oxygen desaturation, hypoglycemia, hypotonia, apnea, lethargy or difficulty arousing, hypertonia or irritability, temperature instability, bradycardia or tachycardia, seizures or seizure-like activity, poor feeding or emesis, hyperbilirubinemia, death before NICU admission.
Time Frame: Birth to first 48 hours of life.
Population: Neonates with admission disposition status
Measure: Count of Participants; unit: Participants
Groups:
- Umbilical Cord Milking - Neonate: Umbilical Cord Milking: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping - Neonate: Early Cord Clamping: The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 872 | 858
Participants
  Total number of neonates admitted to the neonatal intensive care unit for predefined criteria | 199 | 239
  Total number of neonates admitted to neonatal intensive care unit for other criteria | 53 | 52
  Total number of neonates without a neonatal intensive care unit admission | 620 | 567
Statistical Analysis 1: Comparison: Umbilical Cord Milking - Neonate vs Early Cord Clamping - Neonate; Test type: Superiority; p = .87, Hierarchical generalized linear mixed mo; Hierarchical generalized linear mixed models; Least squares mean difference = -0.49, 95% CI 2-sided [-6.36 to 5.37]

2. Secondary Outcome: Median Neonatal Hemoglobin Between 12 to 48 Hours of Life
Description: Single hemoglobin measurement for the neonate which was obtained between 12 to 48 hours of life collected with written consent or as part of standard care.
Time Frame: 12-48 hours of life
Population: Neonates with a hemoglobin measurement obtained between 12 to 48 hours of life either by standard or care of with parental consent.
Measure: Median (Inter-Quartile Range); unit: g/dL
Groups:
- Umbilical Cord Milking - Neonates: Umbilical Cord Milking: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping - Neonates: Early Cord Clamping: The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 298 | 382
g/dL | 18.0 [16.3 to 19.4] | 17.3 [15.7 to 18.8]

3. Secondary Outcome: Number of Neonates Treated With Therapeutic Hypothermia ("Cooling")
Description: Number of neonates that were treated with therapeutic hypothermia (Cooling to 33.5 degrees Celsius) for 72 hours and initiated within the first 6 hours of life.
Time Frame: Birth to 78 hours of life.
Population: Neonates with admission disposition status
Measure: Count of Participants; unit: Participants
Groups:
- Early Cord Clamping - Neonates: Early Cord Clamping: The umbilical cord is clamped as soon as possible within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 829 | 806
Participants | 21 | 35

4. Secondary Outcome: Number of Neonates Treated With Normal Saline Bolus in the First 24 Hours of Life
Description: Number of neonates treated with normal saline bolus in the first 24 hours of life to support blood pressure.
Time Frame: Birth through 24 hours of life
Population: Neonates with admission disposition status
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 823 | 790
Participants | 58 | 56

5. Secondary Outcome: Median Peak Total Serum Bilirubin in Neonates
Description: Highest single measurement of total serum bilirubin obtained as part of standard care to assess hyperbilirubinemia in neonate.
Time Frame: First week of life
Population: All neonates with a total serum bilirubin result from a blood test obtained as part of standard care.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 370 | 450
mg/dL | 8.4 [5.9 to 11.5] | 7 [5.5 to 10.1]

6. Secondary Outcome: Median Transcutaneous Bilirubin in Neonates
Description: Highest single measurement of transcutaneous bilirubin obtained as part of standard care to assess hyperbilirubinemia in each neonate.
Time Frame: birth to 7 days of life
Population: All neonates with a transcutaneous bilirubin measurement in the first week of life as part of standard care.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 393 | 319
mg/dL | 7.1 [5.2 to 9.5] | 6.5 [4.7 to 8.8]

7. Secondary Outcome: Number of Neonatal Deaths
Description: Number of neonatal deaths prior to discharge
Time Frame: Birth to discharge, assessed up to 180 days of life.
Population: Neonates with discharge status available
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 872 | 858
Participants | 0 | 4

8. Other Pre Specified Outcome: Number of Neonates Diagnosed With Mild, Moderate or Severe Hypoxic Ischemic Encephalopathy
Description: Number of neonates with a diagnosis of mild, moderate or severe hypoxic ischemic encephalopathy during neonatal intensive care unit admission.
Time Frame: Birth to discharge, up to 120 days of life.
Population: Neonates with admission disposition status
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 828 | 806
Participants
  Neonates with a diagnosis of mild hypoxic ischemic encephalopathy | 15 | 14
  Neonates with a diagnosis of moderate hypoxic ischemic encephalopathy | 8 | 19
  Neonates with a diagnosis of severe hypoxic ischemic encephalopathy | 4 | 5
  Neonates with no hypoxic ischemic encephalopathy diagnosis | 801 | 768

9. Other Pre Specified Outcome: Median Length of Neonate's Hospitalization in Days Among Participants Discharged Alive
Description: Number of days neonate was admitted to the neonatal intensive care unit from birth to discharge home.
Time Frame: birth to discharge, up to 120 days of life.
Population: Neonates with discharge status
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Early Cord Clamping - Neonates: Early Cord Clamping: The umbilical cord is clamped as early as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 606 | 613
days | 3 [3 to 5] | 3 [3 to 4]

10. Other Pre Specified Outcome: Median Neonatal Admission Blood Pressure
Description: First single neonatal blood pressure measurement by cuff or arterial line obtained on admission to the neonatal intensive care unit and by 48 hours of life.
Time Frame: Birth to 48 hours of life.
Population: Neonates admitted to the neonatal intensive care unit with a blood pressure measurement in the first 48 hours of life.
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Umbilical Cord Milking - Neonates | Early Cord Clamping - Neonates
Number analyzed (Participants) | 182 | 196
mm Hg | 48 [43 to 56] | 46 [41 to 54]

11. Other Pre Specified Outcome: Number of Neonates With Any Cardiorespiratory Support Intervention at Birth
Description: Neonates were assessed for poor tone, poor color (pale, dusky, cyanotic) and poor breathing effort by obstetric provider as part of standard care. Resuscitation assessment and interventions were conducted by neonatal intensive care clinical team. Recorded resuscitation interventions included: use of supplemental oxygen, continuous positive airway pressure respiratory support, positive pressure ventilation respiratory support, endotracheal intubation, chest compressions, epinephrine, normal saline bolus and other cardiorespiratory support medications. Resuscitation interventions including cardiorespiratory support were determined by individual site's clinical standards.
Time Frame: Birth to first hour of life.
Population: Neonates with resuscitation intervention data collected at the time of birth.
Measure: Count of Participants; unit: Participants
Groups:
- Umbilical Cord Milking - Neonatal: Umbilical Cord Milking: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping - Neonatal: Early Cord Clamping: The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Neonatal | Early Cord Clamping - Neonatal
Number analyzed (Participants) | 758 | 730
Participants
  Number of neonates who received supplemental oxygen support in the delivery room | 267 | 337
  Number of neonates who received continuous positive airway pressure support in the delivery room | 295 | 305
  Number of neonates who received positive pressure ventilation support in the delivery room | 313 | 377
  Number of neonates who received endotracheal intubation in the delivery room | 26 | 35
  Number of neonates who received chest compressions in the delivery room | 9 | 7
  Number of neonates administered epinephrine, fluid bolus or other medication in the delivery room | 2 | 3
  Number of neonates with no cardiorespiratory support in the delivery room | 298 | 216

ADVERSE EVENTS:
Time Frame: Neonate's birth to discharge home up to 180 days
Description: Adverse events were assessed for neonates only and were collected from delivery to discharge home.
  Adverse events occurring after discharge were collected as part of follow-up sub-study and will be reported with developmental outcome results is separate publication.
Groups:
- Umbilical Cord Milking-Neonates: All neonates who received umbilical cord milking intervention at the time of birth.
  Umbilical Cord Milking: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping-Neonates: All neonates who received early cord clamping at the time of birth. Early Cord Clamping: The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking-Neonates | Early Cord Clamping-Neonates
All-Cause Mortality (participants affected / at risk) | 0/872 | 4/858
Serious Adverse Events (participants affected / at risk) | 1/872 | 2/858
Other Adverse Events (participants affected / at risk) | 4/872 | 2/858
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Milking-Neonates (N=872) | Early Cord Clamping-Neonates (N=858)
Neonates with intraventricular hemorrhage grade 3 or 4 as assessed by head ultrasound or MRI (Nervous system disorders) | 1 (1) | 2 (2) — Evaluated in neonates admitted to the neonatal intensive care unit and assessed from birth to discharge home, up to 120 days of life.
Neonates with polycythemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — Single hematocrit measurement greater than 65% in the neonate's ﬁrst week of life and assessed from birth to discharge home, up to 120 days of life.
Neonates with pulmonary hemorrhage (Vascular disorders) | 0 (0) | 0 (0) — Evaluated in neonates admitted to the neonatal intensive care unit and assessed from birth to discharge home, up to 120 days of life.
Neonates with hyperbilirubinemia requiring an exchange transfusion (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — Evaluated in neonates admitted to the neonatal intensive care unit and assessed from birth to discharge home, up to 120 days of life.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Milking-Neonates (N=872) | Early Cord Clamping-Neonates (N=858)
Neonates with intraventricular hemorrhage grade 1 (Nervous system disorders) | 3 (3) | 2 (2) — Number of neonates diagnosed with intraventricular hemorrhage grade 1. Assessed from birth to discharge home, up to 120 days of life.
Neonates with intraventricular hemorrhage grade 2 (Nervous system disorders) | 1 (1) | 0 (0) — Number of neonates diagnosed with intraventricular hemorrhage grade 2. Assessed from birth to discharge home, up to 120 days of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT03631940/Prot_SAP_000.pdf